CLINICAL TRIAL: NCT01053169
Title: Non-interventional Observational Study of Beriplex® P/N in Prophylaxis and Treatment of Acute Bleeding Perioperatively (Diagnostic Intervention or Surgery)
Brief Title: Observational Study of Prophylaxis and Treatment of Acute Perioperative Bleeding With Beriplex® P/N (Probe Study)
Status: Completed | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: BE1116_5001; 1492 (Other: CSL Behring)
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Coagulation Protein Disorders; Blood Loss, Surgical; Perioperative Care
Keywords: Coagulopathy; Perioperative bleeding; Prothrombin complex; Liver disease
MeSH Terms: conditions — Coagulation Protein Disorders; Blood Loss, Surgical; Hemostatic Disorders; Liver Diseases | interventions — Factor IX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prophylaxis Cohort: Patients with coagulopathy due to liver disease or other condition requiring correction of coagulopathy who require surgical or diagnostic intervention
  Interventions: Biological: Beriplex® P/N; Biological: Fresh Frozen Plasma (FFP) and Beriplex® P/N; Other: Fresh Frozen Plasma
- Treatment Cohort: Patients experiencing acute bleeding perioperatively
  Interventions: Biological: Beriplex® P/N; Biological: Fresh Frozen Plasma (FFP) and Beriplex® P/N; Other: Fresh Frozen Plasma

INTERVENTIONS:
Biological: Beriplex® P/N — Intravenous infusion, the dosage and the frequency of administration is calculated on an individual patient basis.
  Other Names: Prothrombin complex concentrate
Biological: Fresh Frozen Plasma (FFP) and Beriplex® P/N — FFP is administered before Beriplex® P/N. Each treatment is given as an intravenous infusion, with the dosage of each calculated on an individual patient basis.
  Other Names: Prothrombin Complex Concentrate
Other: Fresh Frozen Plasma — Intravenous infusion, the dosage and the frequency of administration is calculated on an individual patient basis.

SUMMARY:
Beriplex® P/N is made from human plasma (the liquid part of the blood) and contains the coagulation factors II, VII, IX and X which are important for blood clotting (coagulation). Lack of any of these factors means that blood does not clot as quickly as it should and so there is an increased tendency to bleed. This observational study was designed to evaluate the effectiveness of Beriplex® P/N in the prevention (prophylaxis) and treatment of bleeding during surgery (perioperative bleeding) in a routine clinical setting.

ELIGIBILITY:
Inclusion Criteria (All):

For all cohorts:

•≥ 16 years of age

* Received treatment with:

  * Beriplex® P/N
  * or FFP and Beriplex® P/N (in subsequent order)
  * or FFP only
* INR and/or PT results available in connection with administration of Beriplex® P/N or FFP:

  * within 3 hours directly before and after administration of Beriplex® P/N or FFP

In case of Beriplex® P/N use subsequent to FFP, additional results of INR and PT between the administration of the two products

Cohort P (Prophylaxis Group):

* Chronic liver disease, acute liver failure, or other conditions requiring correction of coagulopathy
* Coagulopathy (INR > 1.4 and/or PT ≥ 3 sec of upper limit of normal [ULN])
* Any planned major or minimally invasive procedure, except liver transplantation

Cohort T (Treatment Group):

* Acute perioperative bleeding (as assessed by the investigator)

Exclusion Criteria:

* Treatment with prothrombin complex concentrates (PCCs) other than Beriplex® P/N
* Acquired deficiency of the vitamin K-dependent coagulation factors (e.g., as induced by treatment with oral vitamin K antagonists)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with coagulopathy due to liver disease or other conditions requiring correction of coagulopathy who require surgical or diagnostic intervention and patients experiencing acute bleeding perioperatively
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Adequacy of stopping or preventing bleeding | Up to 24 hours after treatment

SECONDARY OUTCOMES:
Transfusions required | Up to 24 hours after treatment
Clinical trigger for administration of the intervention | Up to 24 hours after treatment
Mortality | Up to 24 hours after treatment
International normalized ratio (INR) | From 3 hours before and up to 24 hours after treatment
Prothrombin time (PT) | From 3 hours before and up to 24 hours after treatment
Receipt of other blood products and /or hemostatic agents | Up to 24 hours after treatment
Vital signs | From 3 hours before and up to 24 hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pratima Chowdary, MRCP, FRCPath, Principal Investigator — The KD Haemophilia Centre & Haemostasis Unit, Royal Free NHS Trust
Locations (6):
- United Kingdom (6):
  - Royal Blackburn Hospital, Blackburn
  - Blackpool, Blackpool
  - Addenbrokes, Cambridge
  - Royal Free Hospital, London
  - Derriford Hospital, Plymouth
  - Southhampton General Hospital, Southhampton